CLINICAL TRIAL: NCT02669082
Title: The Exploratory Study to Investigate the Effect of Ramelteon for Insomnia Patients With Major Depressive Disorder by Using Actigraphy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ramelteon-4002; JapicCTI-163143 (Registry Identifier: JapicCTI); U1111-1177-4116 (Other: WHO)
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Insomnia; Major Depressive Disorder
Keywords: Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major | interventions — ramelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ramelteon 8 mg (Experimental): Ramelteon 8 mg, tablet, orally, once daily at bedtime for 8 weeks.
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Ramelteon — Ramelteon tablets
  Other Names: Rozerem; TAK-375

SUMMARY:
The purpose of this study is to investigate exploratorily the effect of ramelteon 8 mg once daily for 8 weeks in the treatment of insomnia patients with depression by using actigraphy.

DETAILED DESCRIPTION:
The drug being tested in this study is called ramelteon. Ramelteon is being tested to treat people who have insomnia with depression. This study will look at sleep activity of participants who take ramelteon.

The study will enroll approximately 30 patients. Participants will be administered:

• Ramelteon 8 mg

Participants will be asked to take 1 tablet orally at bedtime. This multi-center study will be conducted in Japan. The overall period to participate in this study is 9 weeks (Run-in period for 1 week and treatment period for 8 weeks). Participants will make multiple visits to clinic including the final visit 8 weeks after the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Has difficulty in initiating sleep at least 3 days per week for at least 4 weeks at the time of informed consent.
2. Has Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5)-defined depression.
3. Man or woman between 20 and 64 years of age, inclusive, at the time of informed consent.
4. Outpatient.
5. Meets either of the following criteria based on the 17-item Hamilton Rating Scale for Depression (HAM-D17) both at the start of the run-in period and the start of the study treatment period: has a score of 2 for "6: Insomnia Early", or has a score of 1 for "6: Insomnia Early" AND a score of at least 3 in total for "7: Insomnia Middle" and "8: Insomnia Late".
6. Has a total HAM-D17 score of 16 or under both at the start of the run-in period and the start of the study treatment period.
7. Under treatment of the same antidepressant agents on a stable dose for at least 4 weeks before the start of the run-in period.
8. Goes to bed routinely in a daily life (time for bed between 21.00 p.m. and 1.00 a.m. at least 4 days per week).
9. Actigraphy shows at least 3 days with sleep latency 30 minutes or longer AND total nocturnal sleep time 6.5 hours or shorter on the same day during the run-in period.
10. In the opinion of the principal investigator or investigator, is capable of understanding the contents of the study and complying with study requirements.
11. Is capable of signing and dating the informed consent form in person before any study procedures.

Exclusion Criteria:

1. Has a history of hypersensitivity to ramelteon and melatonin.
2. Has severe liver disorder.
3. Took ramelteon within 4 weeks before the informed consent.
4. Using any insomnia medications (including investigational drugs and unapproved drugs) for 2 weeks before the treatment period.
5. Shift worker or night worker.
6. Has complications of psychiatric or neurological diseases that affect sleep state other than depression.
7. Has a HAM-D17 score of at least 1 for"11: Suicide" at the start of the run-in period or the start of the study treatment period, or any suicide attempts within 24 weeks before or during the run-in period.
8. Pregnant woman, nursing mother, or woman who plans to become pregnant or donate eggs before the informed consent, during the study period or within 4 weeks after the end of the study.
9. Is participating in any other investigational or post-marketing clinical trial/study.
10. For other reason, judged not appropriate for participation in this study by the principal investigator or investigator.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- Japan (7):
  - You Ariyoshi Sleep Clinic, Kitakyushu, Fukuoka
  - Ishikawa Mental Clinic, Sapporo, Hokkaido
  - Minami 1jo Mental Clinic, Sapporo, Hokkaido
  - Senzoku Psychosomatic Clinic, Meguro City, Tokyo
  - Sangenjaya Neurology and Psychosomatic Clinic, Setagaya City, Tokyo
  - Himorogi Kokorono Clinic, Shinjuku, Tokyo
  - Seiwa Hospital, Shinjuku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in Japan from 09 May 2017 to 31 January 2018.
Pre-assignment Details: Participants with a diagnosis of Major Depressive Disorder (MDD) with Insomnia were enrolled in 1 treatment arm: Ramelteon 8 mg.
Period: Overall Study
Arm/Group | Ramelteon 8 mg
Started | 26
Completed | 25
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) was defined as all participants given at least 1 dose of study drug.
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 26
Height [Mean (Standard Deviation); unit: cm] | 168.7 (8.53)
Weight [Mean (Standard Deviation); unit: kg] | 71.08 (12.548)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI)=weight (kg)/[height (m)^2]
  kg/m^2 | 24.94 (3.888)
Smoking Classification [Count of Participants; unit: Participants]
  Non-smoking | 15
  Less than 20 Cigarettes per day | 11
Alcohol Consumption Per Week [Count of Participants; unit: Participants]
  0 day | 13
  1 to 2 days | 8
  3 to 5 days | 3
  6 to 7 days | 2
Duration of Insomnia [Mean (Standard Deviation); unit: years] — Mean duration between the first diagnosis of insomnia and the start of the study was reported.
  years | 4.586 (5.3492)
Duration of Depression [Mean (Standard Deviation); unit: years] — Mean duration between the first diagnosis of depression and the start of the study was reported.
  years | 3.622 (4.5821)
Sleep Latency by Actigraphy [Mean (Standard Deviation); unit: minutes] — Sleep latency was defined as time period measured from "lights out," or bedtime, to the beginning of sleep. Sleep latency was assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep.
  minutes | 44.81 (20.290)
Sleep Latency by Sleep Diary [Mean (Standard Deviation); unit: minutes] — Sleep latency was defined as time period measured from "lights out," or bedtime, to the beginning of sleep. Sleep latency was recorded by the participant in a diary.
  minutes | 51.21 (51.957)
Total Nocturnal Sleep Time by Actigraphy [Mean (Standard Deviation); unit: minutes] — Total nocturnal sleep time was assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep. Total nocturnal sleep time by actigraphy was total time in bed from which sleep latency, nocturnal wake time, and the time from waking up to leaving the bed were subtracted.
  minutes | 314.89 (74.285)
Total Nocturnal Sleep Time by Sleep Diary [Mean (Standard Deviation); unit: minutes] — Total nocturnal sleep time by diary was calculated as total time in bed (awaking hour - bedtime hour) from which sleep latency was subtracted.
  minutes | 407.98 (72.153)
Number of Nocturnal Awakenings by Actigraphy [Mean (Standard Deviation); unit: nocturnal awakenings] — The number of nocturnal awakenings were assessed by actigraphy which is a non-intrusive tool that measures an individual's movement during sleep.
  nocturnal awakenings | 6.05 (2.623)
Number of Nocturnal Awakenings by Sleep Diary [Mean (Standard Deviation); unit: nocturnal awakenings] — The number of nocturnal awakenings were recorded by the participant in a diary.
  nocturnal awakenings | 1.87 (1.079)
Nocturnal Wake Time by Actigraphy [Mean (Standard Deviation); unit: minutes] — Nocturnal wake time is the total time that is scored between nocturnal sleep onset and final wake-up. Nocturnal wake time was assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep.
  minutes | 95.37 (57.572)
Sleep Efficiency by Actigraphy [Mean (Standard Deviation); unit: percentage of sleep] — Sleep efficiency was defined as percentage of sleep in the period potentially filled by sleep-ratio of total sleep time to time in bed calculated as [(Total sleep time/total time in bed) * 100]. Sleep efficiency was assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep.
  percentage of sleep | 67.039 (12.0067)
Daytime Activity Level by Actigraphy [Mean (Standard Deviation); unit: steps] — Daytime activity level, as evaluated by the number of footsteps, was assessed by actigraphy, a non-intrusive tool that measures an individual's movement.
  steps | 5815.17 (2826.252)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Actigraphy-Measured Sleep Latency at the End of the Treatment Period
Description: Sleep latency was defined as time period measured from "lights out," or bedtime, to the beginning of sleep. Sleep latency was assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep. Mean value from the past 7 days was evaluated. A negative change from Baseline indicates improvement.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: Full Analysis Set (FAS) was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
minutes | -6.81 (32.498)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.2955, t-test, 2 sided

2. Secondary Outcome: Change From Baseline in Diary-Measured Sleep Latency at the End of the Treatment Period
Description: Sleep latency was defined as time period measured from "lights out," or bedtime, to the beginning of sleep. Sleep latency was recorded by the participant in a diary. Mean value from the past 7 days at each timepoint was evaluated. A negative change from Baseline indicates improvement.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: FAS was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
minutes | -11.51 (38.087)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.1358, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Actigraphy-Measured Total Nocturnal Sleep Time at the End of the Treatment Period
Description: Total nocturnal sleep time was assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep. Total nocturnal sleep time by actigraphy was total time in bed from which sleep latency, nocturnal wake time, and the time from waking up to leaving the bed were subtracted. Mean value from the past 7 days at each timepoint was evaluated. A positive change from Baseline indicates improvement.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: FAS was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
minutes | 24.20 (87.470)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.1706, t-test, 2 sided; Median

4. Secondary Outcome: Change From Baseline in Actigraphy-Measured Nocturnal Wake Time at the End of the Treatment Period
Description: Nocturnal wake time is the total time that is scored between nocturnal sleep onset and final wake-up. Nocturnal wake time was assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep. Mean value from the past 7 days at each timepoint was evaluated. A positive change from Baseline indicates a worsening.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: FAS was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
minutes | 10.07 (38.739)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.1969, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Actigraphy-Measured Number of Nocturnal Awakenings at the End of the Treatment Period
Description: The number of nocturnal awakenings were assessed by actigraphy which is a non-intrusive tool that measures an individual's movement during sleep. Mean value from the past 7 days at each time point was evaluated. A positive change from Baseline indicates a worsening.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: FAS was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: nocturnal awakenings
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
nocturnal awakenings | 0.53 (1.338)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.0534, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in Actigraphy-Measured Sleep Efficiency at the End of the Treatment Period
Description: Sleep efficiency was defined as percentage of sleep in the period potentially filled by sleep-ratio of total sleep time to time in bed calculated as [(Total sleep time/total time in bed) * 100]. Sleep efficiency was assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep. Mean value from the past 7 days at each timepoint was evaluated. A positive change from Baseline indicates improvement.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: FAS was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage of sleep
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
percentage of sleep | 1.831 (11.2028)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.4125, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Diary-Measured Total Nocturnal Sleep Time at the End of the Treatment Period
Description: Total nocturnal sleep time by diary was calculated as total time in bed (awaking hour - bedtime hour) from which sleep latency was subtracted. Mean value from the past 7 days at each timepoint was evaluated. A positive change from Baseline indicates improvement.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: FAS was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
minutes | 41.17 (85.969)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.0220, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Diary-Measured Number of Nocturnal Awakenings at the End of the Treatment Period
Description: The number of nocturnal awakenings were recorded by the participant in a diary. Mean value from the past 7 days at each timepoint was evaluated. A negative change from Baseline indicates improvement.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: FAS was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: nocturnal awakenings
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
nocturnal awakenings | -0.44 (1.046)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.0420, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Actigraphy-Measured Daytime Activity Level, as Evaluated by the Number of Footsteps, at the End of the Treatment Period
Description: Daytime activity level, as evaluated by the number of footsteps, were assessed by actigraphy, a non-intrusive tool that measures an individual's movement. Mean value from the past 7 days at each timepoint was evaluated. A positive change from Baseline indicates improvement.
Time Frame: Baseline and the end of the Treatment Period (up to Week 8)
Population: FAS was defined as all participants given at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Ramelteon 8 mg
Number analyzed (Participants) | 26
steps | 111.11 (2418.187)
Statistical Analysis 1: Comparison: Ramelteon 8 mg; Data at Baseline compared to the data at the end of the Treatment Period; Test type: Other; p = 0.8166, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to Week 8
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ramelteon 8 mg
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 9/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ramelteon 8 mg (N=26)
Viral upper respiratory tract infections (Infections and infestations) | 5
Somnolence (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT02669082/SAP_000.pdf
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT02669082/Prot_001.pdf